CLINICAL TRIAL: NCT06504472
Title: A Randomized Triple-Blind Placebo-Controlled Study to Evaluate the Effects of a Supplement on Lower Urinary Tract Symptoms in Men.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optimale (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20405
Record Dates: First submitted 2024-07-11; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia; Erectile Dysfunction
Keywords: Pumpkin Seed Extract; Lycopene; Stinging Nettle; Beta-Sitosterols
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia; Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (ProstaThrive™) (Experimental): Participants will take three capsules daily after the final meal of the day for 90 days.
  Interventions: Dietary Supplement: ProstaThrive™ Supplement
- Placebo (Placebo Comparator): Participants will take three placebo capsules daily after the final meal of the day for 90 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ProstaThrive™ Supplement — Participants in this arm will take three ProstaThrive™ capsules daily after the final meal of the day for 90 days.
  Arms: Intervention (ProstaThrive™)
Dietary Supplement: Placebo — Participants in this arm will take three placebo capsules daily after the final meal of the day for 90 days. The placebo capsules will contain an inert substance that mimics the appearance of the ProstaThrive™ supplement.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effects of the ProstaThrive™ supplement on lower urinary tract symptoms (LUTS) in men. It is a 90-day virtual, randomized, placebo-controlled trial with 80 male participants aged 40 and above. The primary endpoint is the reduction in LUTS, while secondary endpoints include changes in sexual function and performance.

DETAILED DESCRIPTION:
This is a virtual two-arm randomized placebo-controlled clinical trial lasting 90 days. Participants will take the ProstaThrive™ supplement or a placebo daily and complete questionnaires at Baseline, Day 30, Day 60, and Day 90. The study will assess the efficacy of ProstaThrive™ on LUTS such as urinary urgency, nighttime urination frequency, perceived urinary flow, and bladder emptying, as well as secondary outcomes related to sexual function.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 40+
* Experience symptoms such as frequent nighttime urination, incomplete bladder emptying, weak urinary stream, and frequent daytime urination
* Difficulty in getting or maintaining an erection
* Willing to avoid introducing any new products or medications targeting LUTS or erectile dysfunction during the study period

Exclusion Criteria:

* Recent surgeries or invasive treatments
* History of prostate or male reproductive cancers
* Urinary issues caused by neurological conditions
* Previous surgery on the genitals, prostate, bladder, or urethra
* Known allergies to product ingredients
* Diagnosed with chronic health conditions impacting study participation
* Current substance abuse
* Participation in other clinical trials
* Taking medications or supplements targeting LUTS or erectile dysfunction

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Change in Lower Urinary Tract Symptoms (LUTS) | Baseline, Day 30, Day 60, and Day 90
  Measured by urinary urgency, nighttime urination frequency (nocturia), perceived urinary flow, and perceived bladder emptying at Baseline, Day 30, Day 60, and Day 90 via questionnaires, including questions adapted from the International Prostate Symptom Score (IPSS).

SECONDARY OUTCOMES:
Change in Sexual Function and Performance | Baseline, Day 30, Day 60, and Day 90
  Measured by the ability to get and maintain an erection at Baseline, Day 30, Day 60, and Day 90 via study-specific questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No